CLINICAL TRIAL: NCT07002359
Title: Assessment of Laboratory Parameters Along With Jugular Vein and Carotid Artery Diameters on Ultrasound in Patients With Gastrointestinal Bleeding
Brief Title: Assessment of Laboratory Parameters and Imaging Findings in Patients With Gastrointestinal Bleeding
Status: Active, not recruiting | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, DENİZ ERDEM, Doktor, Suleyman Demirel University
Other Study IDs: AIBU-ACİL-DE-01
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
METHODS 1.1. Study Design This prospective, cross-sectional, observational study was conducted in the Emergency Department of Süleyman Demirel University Hospital (Isparta, Turkey). From 55,328 annual adult ED admissions, 238 eligible gastrointestinal bleeding (GIB) patients were identified, with 76 enrolled after exclusions. Written informed consent was obtained, and the study is registered at ClinicalTrials.gov.

1.2. Participants Adult patients (≥18 years) with GIB who underwent bedside ultrasonography (May 2023-June 2025) were included. Exclusions: pregnancy, trauma, advanced organ failure, malignancy, inability to consent, or refusal.

Flow Chart:

Suspected GIB: 420

Excluded (no confirmed GIB): 182

Enrolled (confirmed GIB): 238

Included (met criteria): 76

Excluded: 162 (age <18, pregnancy, trauma, comorbidities, no consent, refused hospitalization).

1.3. Sample Size Based on pilot data (effect size 0.5, power 95%, α=0.05), 70 participants were required for significance.

1.4. Data Collection Demographics, labs (Hb, Hct, lactate), hemodynamics (BP, HR, MAP), and outcomes (transfusion, ICU admission, mortality) were recorded.

Ultrasonography: Performed by a certified resident (3 years' experience) using a Terason Usmart 3200T (7.5 MHz probe). IJV and CCA measurements were taken at the thyroid cartilage level.

Scoring: Glasgow-Blatchford score (GBS) assessed bleeding severity.

1.5. Ethical Approval Approved by the local ethics committee (Decision #12, Meeting 92; Feb 20, 2025).

1.6. Quality Evaluation Conducted per Declaration of Helsinki and STROBE guidelines.

1.7. Statistical Analysis Normality: Kolmogorov-Smirnov test.

Comparisons: T-test/Mann-Whitney U (2 groups), ANOVA/Kruskal-Wallis (≥3 groups), Chi-square/Fisher's exact test (categorical).

Correlation: Pearson (GBS vs. US measurements).

Predictive performance: ROC curves (AUC, Youden's Index for cut-offs).

Survival analysis: Kaplan-Meier, Cox regression.

Software: SPSS 27.0, MedCalc® 20.218.

Significance: p < 0.05.

Abbreviations (GIB: Gastrointestinal Bleeding, ED: Emergency Department, ICU: Intensive Care Unit, Hb: Hemoglobin, Hct: Hematokrit, Plt: Platelet, MAP: Mean Arterial Pressure, GBS: Glasgow-Blatchford Score, IJV: Internal Jugular Vein, CCA: Common Carotid Artery, ROC: Receiver Operating Characteristic, AUC: Area Under the Curve, ANOVA: Analysis of Variance, SPSS: Statistical Package for the Social Sciences, STROBE: Strengthening the Reporting of Observational Studies in Epidemiology)

ELIGIBILITY:
Inclusion Criteria: Adult patients aged 18 years and older who presented to the emergency department.

Patients presenting with suspected gastrointestinal bleeding and diagnosed with GIB based on clinical, laboratory, or imaging findings.

Patients who underwent bedside ultrasonography.

Patients who signed the informed consent form (if required).

Patients diagnosed with either upper or lower gastrointestinal bleeding.

Exclusion Criteria:Age <18 years

* Pregnancy
* Trauma-related bleeding
* Chronic comorbidities
* Lack of informed consent
* Refused hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to the emergency department with suspected gastrointestinal bleeding were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Mortality Among Patients with Gastrointestinal Hemorrhage | One Mounth

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi Tıp Fakültesi, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No